CLINICAL TRIAL: NCT05279443
Title: Effect of Yoga-based Exercises on Functional Capacity, Dyspnea, Quality of Life, Depression, Anxiety and Sleep of Healthcare Workers During COVID-19 Pandemic: Prospective Clinical Trial
Brief Title: Effect of Yoga-based Exercises of Healthcare Workers During COVID-19 Pandemic: Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Refiye Önal, MD, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Refiye000000000000000000000001
Record Dates: First submitted 2022-03-13; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pandemic; Yoga; Exercise Therapy; Mind-Body Therapies; Muscle Stretching Exercises
Keywords: yoga; COVID-19; quality of life; healthcare workers; sleep quality
MeSH Terms: conditions — COVID-19; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- yoga-based exercises (Experimental)
  Interventions: Other: yoga-based exercises therapy

INTERVENTIONS:
Other: yoga-based exercises therapy — Accompanied by a certified yoga instructor, and under the supervision of an PMR specialist and a Sports Medicine specialist, YBEs were administered to our patients included in the study for 8 weeks, 2 sessions a week, and with sessions of 60 minutes, using personal mats and equipment in a 2475 m3 (18mx25mx5.5m) gym area that belonged to our hospital, in the form of group therapy for 5 (five) people and in accordance with the social distancing rules. The exercises program was applied as a exercise program consisting of physical postures (asana) to improve the body's muscle strength and flexibility, breathing exercises (pranayama) to increase respiratory function, and relaxation and meditation (dhyana) techniques.

SUMMARY:
To investigate the effect of yoga-based exercises therapy on functional capacity, dyspnea, quality of life, depression, anxiety, and sleep quality in healthcare professionals following COVID-19.

DETAILED DESCRIPTION:
Twenty-six healthcare professionals who were diagnosed with COVID-19, whose treatments were completed, and who were actively working during the subacute period with ongoing complaints were included in the study. The exercises program consisting of stretching, relaxation, isometric strengthening, breathing, and meditation exercises were given to the healthcare professionals under a 60-minute yoga-based exercises program held twice a week for a period of eight weeks. Flexibility and muscle strength measurements of the patients were calculated by the sit and reach test, shoulder flexibility test, and a hand dynamometer. Functional capacity was evaluated with the 6-minute walk test (6MWT), physical activity and dyspnea severity with the modified Medical Research Council (mMRC) dyspnea scale, depression and anxiety level with the Beck Depression and Anxiety Inventory, the quality of life with the SF-36, and sleep quality with the Pittsburgh Sleep Quality Index (PSQI).

ELIGIBILITY:
Inclusion Criteria:prospective clinical trial patients who were COVID-19 PCR (+) and/or diagnosed with COVID-19 pneumonia by computed tomography, completed their medical treatment, had ongoing fatigue, dyspnea, decreased stamina, difficulty in activities of daily living, anxiety, and depression complaints, had an event duration of 2 to 6 months, were actively working (between 25-60 years of age), and had a stable general condition and cognitive ability were included in our study.

Exclusion Criteria:Patients who were hemodynamically unstable, whose cardiac and pulmonary system stability could not be maintained, who had rheumatic, neurological, and psychological disorders, and those who could not continue the program due to working conditions were determined as exclusion criteria.

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | eight week
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity
modified Medical Research Council (mMRC) dyspnoea scale | eight week
  The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing

SECONDARY OUTCOMES:
Beck Anxiety Inventory | eight week
  The BAI is a self-report questionnaire measuring 21 common somatic and cognitive symptoms of anxiety. In a study of adults age 55 years and older in a community-based outpatient facility, the BAI was found to have good discriminant validity

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided